CLINICAL TRIAL: NCT04173039
Title: Diagnostic Value of Antibodies Against Carbamylated Proteins in Psoriatic Arthritis.
Brief Title: Anti-Carbamylated Protein Antibodies in Psoriatic Arthritis
Acronym: CARPAPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Association pour la Recherche Clinique et Immunologique (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 18071A0003
Record Dates: First submitted 2019-11-20; First posted 2019-11-21 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Psoriasis; Arthritis, Psoriatic
MeSH Terms: conditions — Psoriasis; Arthritis, Psoriatic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Controls (Other): Patients with psoriasis and without psoriatic arthritis.
  Interventions: Diagnostic Test: Serum anti-CarP antibodies detection
- Cases (Other): Patients with psoriatic arthritis and with personal or familial psoriasis.
  Interventions: Diagnostic Test: Serum anti-CarP antibodies detection

INTERVENTIONS:
Diagnostic Test: Serum anti-CarP antibodies detection — Serum anti-CarP antibodies detection using an enzyme-linked immunosorbent assay (ELISA) from Inova Diagnostics.

SUMMARY:
Anti-carbamylated protein (anti-CarP) antibodies are present in approximately one-fourth of the patients who are seronegative for both rheumatoid factor and anti-citrullinated protein antibody and who may therefore have psoriatic arthritis. The investigators hypothesized that detection of anti-CarP antibodies in serum may be useful for diagnosis of psoriatic arthritis.

ELIGIBILITY:
Inclusion Criteria:

* "Controls" : Patients with a psoriasis confirmed by a dermatologist and with absence of psoriatic arthritis confirmed by a rheumatologist.
* "Cases" : Patients with psoriatic arthritis fulfilling the classification criteria for psoriatic arthritis (CASPAR), with a diagnosis confirmed by a rheumatologist and associated with personal or familial psoriasis.

Exclusion Criteria:

* "Controls": Presence of any chronic rheumatic inflammatory disease such as psoriatic arthritis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2019-04-24 (Actual); Study Completion 2019-04-24 (Actual)

PRIMARY OUTCOMES:
Sensitivity of anti-carbamylated protein antibodies for the diagnosis of psoriatic arthritis in the psoriatic population | Anti-CarP antibodies will be assessed in the sera collected at the recruitment visit

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Lyon Sud, Pierre-Bénite, France